CLINICAL TRIAL: NCT03250182
Title: A Study to Assess the Pharmacokinetics and Safety of PT010 in Subjects With Moderate to Severe COPD Following Single and Repeat Dose Administration
Brief Title: A Study to Assess the PK and Safety of PT010 in Subjects With COPD Following Single and Repeat Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT010018
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PT010 (Experimental): PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol per protocol. Administered as 2 inhalations per use as instructed in the protocol.
  Interventions: Drug: PT010

INTERVENTIONS:
Drug: PT010 — PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol. Administered as 2 inhalations per use as instructed per the protocol.
  Other Names: PT010; Budesonide, Glycopyrrolate, and Formoterol Fumarate Inhalation Aerosol

SUMMARY:
This is a Phase I open-label, single center study to assess the PK and safety of BGF MDI 320/14.4/9.6 µg in subjects with moderate to severe COPD. Pharmacokinetics will be assessed following a single dose administration on the first treatment day (Day 1) and will be assessed again after 7 days of repeat dosing. This study includes a Screening Period of up to 28 days and a single Treatment Period of 8 days. A follow-up phone call will be conducted at least 5 days but no longer than 7 days after the last dose of study drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Given their signed written informed consent to participate.
* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative serum pregnancy test at Visit 1, and agrees to acceptable contraceptive methods used consistently and correctly for the duration of the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS), or other local applicable guidelines.
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Pre-bronchodilator FEV1/FVC ratio must be <0.70 and pre-bronchodilator FEV1 must be ≥50% and <80% predicted normal value calculated using National Health and Nutrition Examination Survey (NHANES) III reference equations

Key Exclusion Criteria:

* Significant diseases or conditions to : other than COPD, active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, primary pulmonary hypertension, interstitial lung disease and uncontrolled sleep apnea .
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have a history of hypersensitivity to any corticosteroid,
* β2-agonist, muscarinic anticholinergic, or any component of the MDI
* Alpha-1 antitrypsin deficiency as the cause of COPD

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Dorinsky, MD, Study Director — Pearl Therapeutics, Inc.
Locations (1):
- Research Site, Clearwater, Florida, United States

REFERENCES:
- [Derived] Dunn LJ, Kerwin EM, DeAngelis K, Darken P, Gillen M, Dorinsky P. Pharmacokinetics of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler formulated using co-suspension delivery technology after single and chronic dosing in patients with COPD. Pulm Pharmacol Ther. 2020 Feb;60:101873. doi: 10.1016/j.pupt.2019.101873. Epub 2019 Dec 10. PMID 31841699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States from August 2017 to December 2017.
Pre-assignment Details: BGF MDI 320/14.4/9.6 μg oral inhalation as follows:
  * Single-dose on the morning of Day 1 (Visit 3) followed by serial blood draws for 24 hours
  * BID dosing every morning and evening on Day 2 through Day 7 approximately 12 hours apart
  * Single-dose administration on the morning of Day 8 (Visit 5) followed by serial blood draws for 12 hours
Groups:
- PT010: Budesonide, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (BGF MDI) 320/14.4/9.6 µg
Period: Overall Study
Arm/Group | PT010
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects who received at least 1 dose of study drug.
Arm/Group | PT010
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) - Budesonide
Description: Maximum plasma concentration (Cmax) - Budesonide
Time Frame: Day 1
Population: PK Population - All treated subjects who had sufficient data to reliably calculate at least 1 PK parameter for at least one analyte and did not have major protocol deviations which affected the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 29
pg/mL | 709.3 (57.2)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) - Budesonide
Description: Maximum plasma concentration (Cmax) - Budesonide
Time Frame: Day 8 (pre-dose and 2,6,20,40 minutes, 1,2,4,8,10,12 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 27
pg/mL | 663.2 (65.8)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) - Glycopyrronium
Description: Maximum plasma concentration (Cmax) - Glycopyrronium
Time Frame: Day 1 (pre-dose 2,6,20,40 minutes, 1,2,4,8,10,12,18,24 hours post-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 27
pg/mL | 17.2 (80.7)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) - Glycopyrronium
Description: Maximum plasma concentration (Cmax) - Glycopyrronium
Time Frame: Day 8 (pre-dose and 2,6,20,40 minutes, 1,2,4,8,10,12 hours post-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 25
pg/mL | 18.3 (65.4)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) - Formoterol
Description: Maximum plasma concentration (Cmax) - Formoterol
Time Frame: Day 1 (pre-dose 2,6,20,40 minutes, 1,2,4,8,10,12,18,24 hours post-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 29
pg/mL | 6.4 (48.1)

6. Primary Outcome: Maximum Plasma Concentration (Cmax) - Formoterol
Description: Maximum plasma concentration (Cmax) - Formoterol
Time Frame: Day 8 (pre-dose and 2,6,20,40 minutes, 1,2,4,8,10,12 hours post-dose)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 27
pg/mL | 7.4 (38.1)

7. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Budesonide
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Budesonide
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 29
h*pg/mL | 2407.3 (45.4)

8. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Budesonide
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Budesonide
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 27
h*pg/mL | 3004.7 (58.5)

9. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Glycopyrronium
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 22
h*pg/mL | 42.5 (45.8)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Glycopyrronium
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 23
h*pg/mL | 73.9 (52.9)

11. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Formoterol
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Formoterol
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 25
h*pg/mL | 32.6 (30.3)

12. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-12) - Formoterol
Description: Area under the plasma concentration-time curve from 0 to 12 hours (AUC 0-12) - Formoterol
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 25
h*pg/mL | 47.4 (30.0)

13. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-tlast) - Budesonide
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-tlast) - Budesonide
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 29
h*pg/mL | 2731.8 (45.2)

14. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-tlast) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-tlast) - Glycopyrronium
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 27
h*pg/mL | 39.4 (73.5)

15. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC 0-tlast) - Formoterol
Description: Area under the plasma concentration-time curve from 0 to the time of the last measurable plasma concentration (AUC 0-tlast) - Formoterol
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 29
h*pg/mL | 33.4 (43.4)

16. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) - Budesonide
Description: Time to maximum plasma concentration (tmax) - Budesonide
Time Frame: Day 1 (pre-dose 2,6,20,40 minutes, 1,2,4,8,10,12,18,24 hours post-dose), Day 8 (pre-dose and 2,6,20,40 minutes, 1,2,4,8,10,12 hours post-dose)
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PT010
Number analyzed (Participants) | 29
hours
  Day 1 | 0.33 [0.10 to 1.03]
  Day 8: number analyzed (Participants) | 27
  Day 8 | 0.67 [0.10 to 2.00]

17. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) - Glycopyrronium
Description: Time to maximum plasma concentration (tmax) - Glycopyrronium
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PT010
Number analyzed (Participants) | 27
hours
  Day 1 | 0.03 [0.03 to 4.00]
  Day 8: number analyzed (Participants) | 25
  Day 8 | 0.10 [0.03 to 1.00]

18. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) - Formoterol
Description: Time to maximum plasma concentration (tmax) - Formoterol
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | PT010
Number analyzed (Participants) | 29
hours
  Day 1 | 0.33 [0.10 to 9.97]
  Day 8: number analyzed (Participants) | 27
  Day 8 | 0.67 [0.03 to 12.00]

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞) - Budesonide
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC0-∞) - Budesonide
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 24
h*pg/mL | 2996.9 (41.0)

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞) - Glycopyrronium
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC0-∞) - Glycopyrronium
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 4
h*pg/mL | 61.2 (85.1)

21. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 Extrapolated to Infinity (AUC0-∞) - Formoterol
Description: Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC0-∞) - Formoterol
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | PT010
Number analyzed (Participants) | 7
h*pg/mL | 46.0 (33.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of administration of the first dose of study drug to the time of the final follow-up telephone call up to approximately 7 weeks.
Description: The Safety Population was defined as all subjects who receive at least 1 dose of study drug.
Arm/Group | PT010
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PT010 (N=30)
Headache (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations that may arise from this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review and approval and to ensure consistency with the policy in this protocol. Pearl Therapeutics will have the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT03250182/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT03250182/SAP_001.pdf